CLINICAL TRIAL: NCT04543825
Title: Usefulness of Cardiopulmonary Exercise Testing for Cardiovascular Risk Estimation and Frailty Assessment in Liver Transplant Candidates
Status: Completed | Type: Observational
Sponsor: Andres Duarte-Rojo (Other)
Responsible Party: Sponsor-Investigator, Andres Duarte-Rojo, Associate Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Other Study IDs: STUDY19100373
Record Dates: First submitted 2020-09-02; First posted 2020-09-10 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Cardiovascular Diseases+Liver Transplantation
Keywords: 6-minute walk test, cirrhosis, frailty, major adverse cardiac event
MeSH Terms: conditions — Fibrosis; Frailty | interventions — Exercise Test

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- CPET: Patients with cirrhosis who have been wait listed for liver transplant or are undergoing liver transplant evaluation and will undergo cardiopulmonary exercise testing (CPET).
  Interventions: Device: Cardiopulmonary exercise testing

INTERVENTIONS:
Device: Cardiopulmonary exercise testing — Subjects will perform cardiopulmonary exercise testing which consists of biking on a cycle ergometer (recumbant stationary bicycle) while breathing through a mouthpiece or mask to measure the oxygen and carbon dioxide in the subject's breath. We will also do impedance cardiography, an FDA-approved test to check how the heart functions during exercise. For this test we will attach 6 electrodes (total) to the chest and back (similar to an EKG), so that we can measure the quantity of blood coming out of the heart on every heartbeat. Each evaluation will also include cardiac testing looking for coronary artery disease (CAD).

SUMMARY:
Patients undergoing liver transplantation (LT) have a high risk for cardiovascular disease (CVD). Frailty is a frequent condition among LT candidates. Together, CVD and frailty are major causes of morbidity and mortality before and after LT. Conventional methods to diagnose and predict CVD in LT candidates lack sensitivity and clinically relevant application. However, cardiopulmonary exercise testing (CPET) can directly estimate coronary artery disease, cirrhotic cardiomyopathy, and indirectly assess frailty. Such versatility of CPET has caused it to become the standard of care in many LT centers outside of the United States.

In preliminary work (funded internally by the Pittsburgh Liver Research Center) that will be used to fund a more definitive study (RO1), the investigators plan to investigate CVD and frailty in LT candidates, both from existing standard of care (SOC) methods and CPET. The investigators expect results to improve the current capacity to assess and prognosticate CVD and frailty in LT, ultimately changing practice.

DETAILED DESCRIPTION:
Patients undergoing liver transplantation (LT) have a high risk for cardiovascular disease (CVD). Frailty is a frequent condition among LT candidates. Together, CVD and frailty are major causes of morbidity and mortality before and after LT. Conventional methods to diagnose and predict CVD in LT candidates lack sensitivity and clinically relevant application. However, cardiopulmonary exercise testing (CPET) can directly estimate coronary artery disease, cirrhotic cardiomyopathy, and indirectly assess frailty. Such versatility of CPET has caused it to become the standard of care in many LT centers outside of the United States. In preliminary work that will be used to fund a more definitive study (RO1), the investigators plan to investigate CVD and frailty in LT candidates, both from existing standard of care (SOC) methods and CPET. The investigators expect results to improve the assessment of CVD and frailty in LT, ultimately changing practice. The investigators' proposal will pursue the following Specific Aims (SA):

Aim 1: Prospectively determine agreement between cardiopulmonary exercise testing and cardiac stress testing, for the identification of subclinical coronary artery disease in liver transplant candidates.

Aim 2: Prospectively determine agreement between cardiopulmonary exercise testing and dobutamine stress echocardiogram (DSE) or impedance cardiography, for the identification of cirrhotic cardiomyopathy in liver transplant candidates.

Aim 3: Prospectively determine agreement between peak oxygen consumption from cardiopulmonary exercise testing and the liver frailty index or the six-minute walk test, for the identification of frailty in liver transplant candidates.

ELIGIBILITY:
Inclusion Criteria:

* Wait listed patients with cirrhosis or those undergoing LT evaluation

Exclusion Criteria:

* Subjects younger than 45 or older than 75 years
* Subjects with platelets <30,000
* Subjects with international normalized range (INR) >3
* Subjects with glomerular filtration rate (GFR) <30
* Subjects with left main artery stenosis
* Subjects with moderate/severe stenotic valvular disease
* Subjects with atrial fibrillation and other arrythmias
* Subjects with resting ventricular ejection fraction <50%
* Subjects with portopulmonary hypertension
* Subjects with severe chronic obstructive pulmonary disease (COPD)
* Subjects with an exercise contraindication

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients waitlisted for a liver transplant or undergoing liver transplant evaluation
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2020-09-25 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Cardiopulmonary exercise testing and cardiac stress testing | 12 months
  Agreement between cardiopulmonary exercise testing and cardiac stress testing, for the identification of subclinical coronary artery disease in liver transplant candidates.
Cardiopulmonary exercise testing and dobutamine stress echocardiogram | 12 months
  Agreement between cardiopulmonary exercise testing and dobutamine stress echocardiogram (DSE) or impedance cardiography, for the identification of cirrhotic cardiomyopathy in liver transplant candidates.
Peak oxygen consumption from cardiopulmonary exercise testing | 12 months
  Agreement between peak oxygen consumption from cardiopulmonary exercise testing and the liver frailty index or the six-minute walk test, for the identification of frailty in liver transplant candidates.

CONTACTS AND LOCATIONS:
Overall Officials: Andres Duarte-Rojo, MD, Principal Investigator — University of Pittsburgh
Locations (2):
- United States (2):
  - Mayo Clinic Arizona, Phoenix, Arizona
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No
The investigators will construct a REDCap database to collect deidentified research data, as per IRB-approved clinical research form, for a combined analysis of all recruiting centers